CLINICAL TRIAL: NCT05983133
Title: A Phase 1 Study of PF-08046052/SGN-EGFRd2 in Advanced Solid Tumors
Brief Title: A Study of PF-08046052/SGN-EGFRd2 in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNEGFRd2-001; C5841001 (Other: Alias Study Number)
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of the Head and Neck; Pancreatic Ductal Adenocarcinoma
Keywords: CRC; Colon Cancer; Rectal Cancer; NSCLC; HNSCC; PDAC; Seattle Genetics
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-08046052/SGN-EGFRd2 (Experimental): PF-08046052/SGN-EGFRd2 monotherapy
  Interventions: Drug: PF-08046052

INTERVENTIONS:
Drug: PF-08046052 — Given into the vein (IV; intravenously)
  Other Names: SGN-EGFRd2

SUMMARY:
This study will test the safety of a drug called PF-08046052/SGN-EGFRd2 in participants with advanced solid tumors. It will also study the side effects of this drug. A side effect is anything a drug does to the body besides treating the disease.

Participants will have cancer that cannot be removed (unresectable) or has spread through the body (metastatic).

This study will have three parts. Parts A and B of the study will find out how much PF-08046052/SGN-EGFRd2 should be given to participants. Part C will use the dose found in parts A and B to find out how safe PF-08046052/SGN-EGFRd2 is and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Tumor types:

  * For Part A: Participants must have disease that is relapsed, refractory, or be intolerant to standard of care therapies, and in the judgement of the investigator must have no appropriate standard therapy available at the time of enrollment. Participants must have histologically- or cytologically confirmed metastatic or unresectable solid malignancy from one of the following tumor types:

    * Colorectal cancer (CRC)
    * Non-small cell lung cancer (NSCLC)
    * Head and neck squamous cell cancer (HNSCC)-non-nasopharyngeal subtype ONLY; nasopharyngeal subtype is not eligible.
  * For Part B: Participants must have disease that is relapsed, refractory, or be intolerant to standard of care therapies, and in the judgement of the investigator must have no appropriate standard therapy available at the time of enrollment.

    * The tumor type(s) to be enrolled in dose optimization will be identified by the sponsor from among those specified in Part A.
  * For Part C: Participants must have disease that is relapsed or refractory or be intolerant to standard of care therapies as specified below, unless contraindicated:

    * CRC

      * Participants must have unresectable locally advanced or metastatic CRC.
      * Prior therapy: Participants must have received prior fluoropyrimidine, oxaliplatin and irinotecan. Participants with defective mismatch repair and microsatellite instability high (dMMR/MSI-H) should have received prior treatment with pembrolizumab, a nivolumab-containing regimen, or other available anti-PD-1 (programmed cell death protein 1) or anti PD L1 (programmed cell death 1 ligand) agents.
    * NSCLC

      * Participants must have unresectable locally advanced or metastatic NSCLC.
      * Prior therapy: Participants must have received platinum-based therapy and at least 1 PD-1/PD-L1 inhibitor. These agents may have been administered either as single agents or in combination. Participants with an activating mutation or rearrangement (eg, EGFR, anaplastic lymphoma kinase [ALK], etc.) must have received available targeted agents if eligible by biomarker status and local standard of care.
    * HNSCC

      * Participants must have unresectable locally advanced or metastatic HNSCC - non-nasopharyngeal subtype ONLY; nasopharyngeal subtype is not eligible.
      * Prior therapy: Participants must have received platinum-based therapy and a PD-1/PD-L1 inhibitor, if eligible by biomarker status and local standard of care. These agents may have been administered either as single agents or in combination.
    * Pancreatic ductal adenocarcinoma (PDAC)

      * Participants must have unresectable locally advanced or metastatic PDAC.
      * Prior therapy: Participants must have received gemcitabine- or FOLFIRINOX-based therapy.
* Participants should provide archival tumor tissue if available and also agree to biopsies, if medically feasible
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Measurable disease at baseline per RECIST 1.1 criteria.

Exclusion Criteria:

* History of another malignancy within 3 years before the first dose of study treatment, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death
* Known active central nervous system metastases or leptomeningeal disease. Participants with previously treated brain metastases may participate provided they are

  * clinically stable for at least 4 weeks prior to study entry after brain metastases treatment,
  * they have no new or enlarging brain metastases,
  * and are off of corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study drug.
* Treatment with an aminobisphosphonate IV (eg ibandronate, pamidronate, zoledronate, etc.) within 4 weeks of the first dose of study treatment.
* Participants with history of thromboembolic phenomena within 6 months prior to the first dose of study intervention, or with contraindication to thromboembolism prophylaxis (if clinically indicated) for a previous history of thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 90 days after last study treatment, up to approximately 1 year
  An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after last study treatment, up to approximately 1 year
Number of participants with dose limiting toxicities (DLTs) | Up to 35 days
Number of participants with DLTs by dose level | Up to 35 days

SECONDARY OUTCOMES:
Number of participants with antidrug antibodies (ADAs) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
Pharmacokinetic (PK) parameter - Area under the curve (AUC) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Time to maximum concentration (Tmax) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Apparent terminal half-life (t1/2) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after last study treatment, up to approximately 1 year
  To be summarized using descriptive statistics
Objective response rate (ORR) | Up to approximately 2 years
  ORR is defined as the proportion of participants with an objective response per Response Evaluation in Solid Tumors (RECIST) 1.1 per investigator. A participant is determined to have an objective response if, based on RECIST 1.1, they achieve a complete response (CR) or partial response (PR) after initiation of treatment and at or prior to the EOT disease assessment.
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per RECIST 1.1 or to death due to any cause, whichever comes first
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from start of SGN-EGFRd2 to first documentation of disease progression or death due to any cause, whichever comes first
Overall survival (OS) | Up to approximately 3 years
  OS is defined as the time from start of SGN-EGFRd2 to date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (22):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Santa Monica UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Moffitt Cancer Center McKinley Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Atrium Health Wake forest Baptist, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center / Wake Forest University, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital, University of Utah, Salt Lake City, Utah
  - Huntsman Cancer Institute, University Of Utah, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
- United Kingdom (2):
  - University College London Hospital, NIHR UCLH Clinical Research Facility, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNEGFRd2-001